CLINICAL TRIAL: NCT00682318
Title: Effects of Fish Oil and Red Wine on Oxidative Stress Biomarkers: a Randomized Double-blinded Trial on the Modulation of the Eicosanoid and Isoprostane Pathways in Healthy Subjects by Omega-3 Polyunsaturated Fatty Acids and Red Wine.
Brief Title: Effects of Fish Oil and Red Wine on Oxidative Stress Biomarkers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carsten Skarke, MD (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Carsten Skarke, MD, Research Assistant Professor of Medicine, Institute for Translational Medicine and Therapeutics, ITMAT, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 807069
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Fish oil; red wine; alcohol; oxidative stress; Healthy volunteers
MeSH Terms: interventions — Fish Oils; Safflower Oil; Ethanol; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil (Experimental): Omega-3 polyunsaturated fatty acids (n-3 PUFA)
  Interventions: Drug: Fish Oil; Dietary Supplement: Ethanol; Dietary Supplement: Omega-3 polyunsaturated fatty acids
- Safflower Oil (Active Comparator): Omega-6 polyunsaturated fatty acids (n-6 PUFA)
  Interventions: Dietary Supplement: Safflower Oil; Dietary Supplement: Ethanol; Dietary Supplement: Omega-6 polyunsaturated fatty acid

INTERVENTIONS:
Drug: Fish Oil — Part 1.1: Dose of 9.3 g/day EPA plus 7.5 g/day DHA;
  Part 2a (run-in phase): Dose of 1 time 2 capsules per day of Lovaza (total of 1.7 g/d ω-3 PUFA consisting of 930 mg/day EPA and 750 mg/day DHA) for 29±1 days;
  Part 2a (study arm): Dose of 3 times 4 capsules per day of Lovaza (total of 10.1 g/d ω-3 PUFA consisting of 5580 mg/day EPA and 4500 mg/day DHA) for 29±1 days
  Other Names: LovazaTM (former name: Omacor®)
  Arms: Fish oil
Dietary Supplement: Safflower Oil — Part 2a: (Study Arm): Omega-6 polyunsaturated fatty acids 3 times 4 capsules per day (total of 10.2 g/d ω-6 PUFA) for 29±1 days
  Other Names: Omega-6 polyunsaturated fatty acids
  Arms: Safflower Oil
Dietary Supplement: Ethanol — Part 1 & Part 1.1:
  Dose of 0.9 g/kg body weight 98% alcohol solution
  Part 2a:
  Doses of 0.4 and 0.9 g/kg body weight 98% alcohol solution and a control placebo drinking solution
  Part 2b, Part 3:
  Doses of 0.4, 0.6 and 0.9 g/kg body weight 98% alcohol solution
Dietary Supplement: Omega-3 polyunsaturated fatty acids — Part 2b:
  Alimentary diet delivering ≈ 500 mg/day EPA/DHA,or Alimentary diet delivering ≈ 900-1000 mg/day EPA/DHA, or Alimentary diet delivering ≈ 1500-1800 mg/day EPA/DHA;
  Part 3:
  Alimentary diet delivering EPA/DHA in a quantity to be determined by Part 2b.
  Other Names: n-3 PUFA alimentary supplementation
  Arms: Fish oil
Dietary Supplement: Omega-6 polyunsaturated fatty acid — Part 2b:
  Control omega-6 fatty acid alimentary diet (<130 mg/day EPA/DHA)
  Other Names: n-6 PUFA alimentary supplementation
  Arms: Safflower Oil

SUMMARY:
The American Heart Association and the American College of Cardiology (AHA/ACC) recently encouraged "increased consumption of omega-3 fatty acids in the form of fish or capsule form (1 g/day) for risk reduction" and stated that "for treatment of elevated triglycerides, higher doses are usually necessary for risk reduction" (Smith SC et al. Circulation 2006;113:2363-72). These recommendations are based on conflicting evidence about the efficacy of the omega-3 treatment with data derived from single randomized trials or non-randomized studies (Smith SC et al. Circulation 2006;113:2363-72). Much effort has been undertaken to elucidate the role of omega-3 fatty acids in the development of cardiovascular disease, but even recent meta-analyses deliver no clear picture; they either favor (Mozaffarian D Jama 2006;296:1885-99) or reject (Hooper L Bmj 2006;332:752-60) the hypothesis of cardioprotective effects of omega-3 FAs.

The objective of the clinical study is to study the effects of fish oil on blood and urinary markers of inflammation and cell stress. By using different permutations of high-dose supplementation of omega-3 and omega-6 fatty acids versus different alimentary omega-3 fish doses and grain alcohol versus different kinds of red wine, this trial will study how omega-3 fatty acids, ethanol and red wine constituents modulate biomarkers of inflammation and cell stress.

DETAILED DESCRIPTION:
This clinical study comprises several parts:

Part 1: Single-arm open oral administration of ethanol in n=40 healthy participants.

Part 1.1: Single-arm open oral administration of fish oil capsules and ethanol in n=12 healthy participants.

Part 2a: Randomized double-blind oral administration of fish oil or safflower oil capsules and ethanol in n=44 healthy participants.

Part 2b: Randomized double-blind oral administration of fish foods or control diet and open oral administration of ethanol in n=40 healthy participants.

Part 3: Randomized double-blind oral administration of fish foods or control diet and red wine beverages in n=40 healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 - 60,
* Subjects must be in good health as based on medical history, physical examination, vital signs, and laboratory tests.
* All Subjects have to adhere to the following criteria:
* Must be non-smoking volunteers (both male and non-pregnant females) due to a significant influence of smoking and overweight on the outcome measures of lipid peroxidation,
* Must be of normal weight with a body mass index (BMI) ≤ 25. The correlation between the BMI number and body fatness is fairly strong; however it varies by sex, race, and age. These variations include the following examples: At the same BMI, women tend to have more body fat than men; at the same BMI, older people, on average, tend to have more body fat than younger adults; highly trained athletes may have a high BMI because of increased muscularity rather than increased body fatness; source at http://www.cdc.gov/healthyweight/assessing/bmi/adult_BMI/index.html. Therefore, subjects with a BMI > 25 can be enrolled at the discretion of the PI in writing.
* Female subjects of child bearing potential must be using a medically acceptable method of contraception (oral contraception, depo-provera injection, IUD, condom with spermicide, diaphragm, cervical cap, progestin implant, abstinence, tubal ligation, oophorectomy, TAH) throughout the entire study period. All female subjects must consent to a urine pregnancy test at screening and just prior to the start of each treatment phase of the study (first study visit, every ethanol administration visit, at first visit of fish oil administration), and during the third week of fish oil administration. All pregnancy tests must be negative at all time points.
* Male subjects must be surgically sterile and/or agree to use condoms throughout the duration of the study.
* Persons who consume vitamin supplements are required to undergo a "washout period" of ≥ five weeks without supplement prior to study enrollment (in analogy to Block G, et al. Am J Epidemiol 2002; 156: 274)
* Urine ethanol assessment indicating abstinence.

Exclusion Criteria:

* Female subjects who are pregnant or nursing a child.
* Subjects, who have received an experimental drug, used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening.
* Subjects with any coagulation, bleeding or blood disorders.
* Subjects with nutritional inefficiencies in Fe, Zn, Cu, Mg (according to 61)
* Subjects who are sensitive or allergic to fish, fish oil or fish-containing products.
* Subjects with any evidence of cancer or history of significant cardiovascular disease (including stroke or TIA), renal, hepatic, respiratory, endocrine, metabolic, hematopoietic or neurological disorder.
* Subjects with a systolic blood pressure above 160 or a diastolic blood pressure above 95,
* Subjects with any evidence of GI disorders that could interfere with fat absorption
* Subjects with an intention to lose weight during their participation in the trial
* Subjects with any abnormal laboratory value or physical finding that according to the investigator may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject. Subjects who have had a history of drug or alcohol abuse within the last 6 months.
* Carbohydrate-deficient transferrin > 6% indicating chronic alcohol abuse
* Complete abstinence from alcohol
* Intake of more than three alcoholic drinks per day
* Subjects with a history of cancer, including skin cancer

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-05 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Urinary isoprostane concentrations | Hours and days
  urinary isoprostanes will be analyzed raw (i.e. untransformed, including the Time factor: Baseline vs Peak)

SECONDARY OUTCOMES:
Urinary eicosanoid concentrations | Hours and days
  Time-dependency of urine eicosanoid and isoprostane formation after acute oral ethanol
Plasma eicosanoid concentrations | Hours and days
  plasma eicosanoid response after a single oral dose of 0.9 g/kg body weight 98% ethanol.
Blood alcohol concentrations | Hours and days
  Evaluation of acute toxic alcohol effects
Blood fatty acid composition | Hours to months
  Oral administration of omega-3 and omega-6 fatty acids
Compositional Changes in the Intestinal Microbiome | Hours and days
  Collection of stool samples

OTHER OUTCOMES:
Metabolomics, Lipidomics, Transcriptomics | Baseline, after low and high doses of fish oil supplementation, after high doses of safflower oil supplementation, after ethanol ingestion
  Exploring potential interactions between polyunsaturated fatty acids and ethanol

CONTACTS AND LOCATIONS:
Overall Officials: Garret A FitzGerald, M.D., Principal Investigator — Institute for Translational Medicine & Therapeutics, School of Medicine; Carsten Skarke, M.D., Principal Investigator — Institute for Translational Medicine & Therapeutics, SOM
Locations (1):
- Institute for Translational Medicine and Therapeutics (ITMAT), University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States